CLINICAL TRIAL: NCT03485885
Title: Bioavailability of Maqui Berry Extracts (Delphinol® / MaquiBright®) in Healthy Subjects
Brief Title: Bioavailability of Maqui Berry Extract (MBE) in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Anklam Extrakt (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: BTS1093/17
Record Dates: First submitted 2018-03-19; First posted 2018-04-03 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Bioavailability
Keywords: anthocyanins, maqui berries, bioavailability
MeSH Terms: interventions — Anthocyanins; Delphinol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maqui Berry Extract (MBE): To be tested for the extracts bioavailability
  Interventions: Dietary Supplement: Standardized maqui berry extract enriched in anthocyanins

INTERVENTIONS:
Dietary Supplement: Standardized maqui berry extract enriched in anthocyanins — Single oral intake of 1000mg standardized maqui berry extract (in 4 capsules - 250mg each) with 200ml still water
  Other Names: Delphinol® / MaquiBright®

SUMMARY:
The aim of the present study is to describe the bioavailability for the proprietary standardized maqui berry extracts Delphinol® and MaquiBright® enriched in anthocyanins and in particular delphinidins. The analyses are based on two selected key substances namely delphinidin-3-glucoside and cyanidin-3-sambubioside and their metabolism to phenolic acids.

The bioavailability of anthocyanins specific for Delphinol®/MaquiBright® was analyzed in plasma sample kinetics (at 0h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h and 8h after intake of 1000mg standardized maqui berry extract in capsules) in 12 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able and willing to sign the Informed Consent Form prior to screening evaluations
2. Sex: female and male
3. Age: 18- 50 years
4. BMI ≥19 or ≤30 kg/m²
5. Non-smoker
6. Subject is in good physical and mental health as established by medical history, physical examination, electrocardiogram, vital signs, results of biochemistry, haematology

Exclusion Criteria:

Subjects who met one or more of the following criteria are not eligible:

1. Relevant history or presence of any medical disorder, potentially interfering with this study (e.g. mal absorption, chronic gastro-intestinal diseases, etc.)
2. For this study clinically relevant abnormal laboratory, ECG, vital signs or physical findings at screening
3. Coffee consumption >3 cups / day
4. Consumption of more than 5 portions fruits and vegetables per day
5. Blood donation within 1 month prior to study start or during study
6. Regular intake of drugs or supplements possibly interfering with this study (e.g. Vitamin C, E, OPC etc.) within 2 weeks prior to study start or during study (Vitamin D with highest dosage of 1000 I.E. per day will be allowed)
7. Vegetarians / vegans
8. Drug-, alcohol- and medication abuses
9. Known HIV-infection
10. Known acute or chronic hepatitis B and C infection
11. Relevant allergy or known hypersensitivity against compounds of the study preparations
12. Known pregnancy, breast feeding or intention to become pregnant during the study
13. Participation in another clinical study within the last 4 weeks and concurrent participation in another clinical study
14. Anticipating any planned changes in lifestyle for the duration of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: normal population
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Quantification of two specific maqui berry anthocyanins: namely Delphinidin-3-O-glucoside and Cyanidin-3-O-sambubioside in a kinetics, evaluating the change between baseline and selected time points (see below). | Kinetics: baseline to 0.5 hours, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours after intake
  Specific anthocyanins related to maqui berry extract (Delphinol® / MaquiBright®) were measured in plasma samples of healthy subjects and assessed as change to baseline. Method: LC-MS/MS (unit [nmol/L]).
Quantification of two specific maqui berry anthocyanin derived metabolites: namely gallic acid and protocatechuic acid in a kinetics, evaluating the change between baseline and selected time points (see below). | Kinetics: baseline to 0.5 hours, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours after intake
  Specific anthocyanin derived metabolites related to maqui berry extract (Delphinol® / MaquiBright®) were measured in plasma samples of healthy subjects and assessed as change to baseline. Method: LC-MS/MS. Results will most probably be assessed as "AUC" (area under the curve).
Ferric reducing ability of plasma (FRAP) measurement in a kinetics, evaluating the change between baseline and selected time points (see below). | Kinetics: baseline to 0.5 hours, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours after intake
  The FRAP assay was performed to assess the "antioxidant power" / "antioxidant capacity" of the plasma after intake of maqui berry extract (Delphinol® / MaquiBright®). Method: photometric / absorption maximum at 593 nm (unit [µmol/l])

CONTACTS AND LOCATIONS:
Locations (1):
- Nutritional CRO & Study site; BioTeSys GmbH, Esslingen am Neckar, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No